CLINICAL TRIAL: NCT06717919
Title: Hypothermic Oxygenated Perfusion (HOPE) Against Cancer Recurrence in HCC Liver Transplantation - International Multicentre Parallel Group Interventional RCT
Brief Title: HOPE Against Cancer Recurrence in HCC
Acronym: HOPE4Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Philipp Dutkowski (Other)
Responsible Party: Sponsor-Investigator, Philipp Dutkowski, Sponsor representative and Principal Investigator, Clarunis - Universitäres Bauchzentrum Basel
Organization: Clarunis - Universitäres Bauchzentrum Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221622
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplantation; HCC; Oncological Outcomes
Keywords: HOPE; randomised controlled trial; multicentre; hepatocellular carcinoma; liver transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional cold storage (Active Comparator): Conventional cold storage at 4°C will be performed with precooled preservation solution according to local standard of care. For cold storage at the Swiss centres, IGL-1 (Institute George Lopez) is used for cold storage. Liver transplant centres in other European countries, use mainly three other storage solutions (Histidine trypophan-ketoglutarat, HTK and University of Wisconsin, UW solution, Celsior) in accordance to their national guidelines.
  Interventions: Procedure: Conventional cold storage
- Hypothermic oxygenated perfusion (Experimental): All study centres will use either VitaSmart, Liver assist or Perlife devices for machine liver perfusion, with a pressure controlled hypothermic oxygenated liver perfusion through the portal vein (HOPE) or through the portal vein and the hepatic artery (DHOPE), targeting a flow rate between 200-250 ml/min at a pressure of 3 mmHg, and a perfusate temperature between 8-12°C. The perfusate consists of 3L re-circulating Belzer MPS® (Bridge to Life Ltd.) with an active oxygenation (70-110 kPa). The minimum perfusion duration is defined at 2 hours, while perfusion is generally continued until the recipient hepatectomy is completed. The perfusion will exclusively be performed in the recipient centre after initial cold storage and bench preparation of the liver for implantation.
  The perfusion devices are routinely used in all participating centres (VitaSmart, Bridge to Life®, Liver Assist, XVIVO®, Perlife, Aferitica®).
  Interventions: Procedure: Hypothermic oxygenated perfusion

INTERVENTIONS:
Procedure: Hypothermic oxygenated perfusion — All study centres will use either VitaSmart, Liver assist or Perlife devices for machine liver perfusion, with a pressure controlled hypothermic oxygenated liver perfusion through the portal vein (HOPE) or through the portal vein and the hepatic artery (DHOPE), targeting a flow rate between 200-250 ml/min at a pressure of 3 mmHg, and a perfusate temperature between 8-12°C. The perfusate consists of 3L re-circulating Belzer MPS® (Bridge to Life Ltd.) with an active oxygenation (70-110 kPa). The minimum perfusion duration is defined at 2 hours, while perfusion is generally continued until the recipient hepatectomy is completed. The perfusion will exclusively be performed in the recipient centre after initial cold storage and bench preparation of the liver for implantation. The perfusion devices are routinely used in all participating centres.
  Arms: Hypothermic oxygenated perfusion
Procedure: Conventional cold storage — Conventional cold storage at 4°C will be performed with precooled preservation solution according to local standard of care. For cold storage at the Swiss centres, IGL-1 (Institute George Lopez) is used for cold storage. Liver transplant centres in other European countries, use mainly three other storage solutions (Histidine trypophan-ketoglutarat, HTK and University of Wisconsin, UW solution, Celsior) in accordance to their national guidelines.
  Arms: Conventional cold storage

SUMMARY:
Liver transplantation is often performed to treat liver cancer, or hepatocellular carcinoma (HCC), in patients with impaired liver function due to cirrhosis. A shortcoming, however, is tumor recurrence after transplantation. Approximately 15 % of patients receiving livers develop recurrence and this depends on the quality of the liver received.

Machine liver perfusion, for example, hypothermic oxygenated liver perfusion (HOPE), which means that the organ is perfused with an oxygen-rich fluid in a cold environment before transplantation, is a novel method to improve the quality of livers before implantation. The standard of care is cold storage without perfusion.

The objective of this study is to compare the survival after tumor recurrence of patients after liver transplantation for HCC between perfused and not perfused livers. This study's hypothesis is that survival without tumor recurrence is improved when the liver is perfused before implantation.

The study involves transplant centers worldwide, and adults with HCC waiting for liver transplantation are included. 220 Patients will be recruited within 12 months and then observed for at least 2 years after transplantation. To provide the most valid results, the patients will be randomly allocated to either the organ perfusion group or a control group with standard-of-care cold storage of the organ.

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients (>18y), listed for liver transplantation with documented HCC (Liver Imaging Reporting and Data System (LIRADS) 5 lesion in magnetic resonance imaging or computer tomography of the liver or biopsy proven),
* within up to seven criteria, i.e. HCC with seven as the sum of the diameter of the largest tumour (in cm) and the number of tumours at the time point of liver transplantation,
* written informed consent for the trial. This also includes patients beyond the up to seven criteria after successful downsizing of the HCC

Exclusion Criteria:

* Donation after circulatory death (DCD) liver grafts
* Combined liver transplants
* Partial liver transplants
* Combined or mixed hepatocellular cholangiocarcinoma (cHCC-CCC) or pure cholangiocarcinoma or other malignancies in histopathology of the liver explant
* Systemic antitumoural medical treatment with checkpoint inhibitors or multikinase inhibitors
* Post-transplant treatment with mTOR inhibitors
* Acute and unexpected medical contraindications
* Pregnancy
* Cold storage time of > 10 hours (both study arms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | 24 months
  Post transplant HCC recurrence free survival, i.e. the time interval a patient is alive without HCC recurrence after transplantation, i.e., until either HCC recurrence is observed, or the patient dies from any cause.

SECONDARY OUTCOMES:
HCC recurrence (while alive) | 24 months
  Number of HCC recurrences
HCC recurrence (while alive) | 24 months
  Time to recurrence of HCC
HCC-related death | 24 months
  Death related to HCC
HCC-related death | 24 months
  Time to HCC related death
Death from any other causes than HCC | 24 months
  Death not related to HCC
Death from any other causes than HCC | 24 months
  Time to death not related to HCC
Mean number of circulating tumour deoxyribonucleic acid (DNA) in blood | 6 months
  This will be measured before transplantation (baseline), at discharge and at 6 months after transplantation. This endpoint will add information on the risk of tumour recurrence by seeding circulating cells.
Mean number of high-mobility-group-protein B1 (HMGB-1) in blood | 1 week
  This will be measured at the time of transplantation (baseline) and 1 week after transplantation.
  This endpoint will add information on danger signalling in both study arms during early and late reperfusion.
Median Rejection Activity Index | 6 months
  The Rejection Activity Index (RAI) in liver histology (biopsy) is performed at 6 months after transplantation. This endpoint assessed in liver histology (biopsy) will show endothelial and T cell activation in implanted livers within the first months after 6 months.
  The RAI can be used to score liver allograft biopsies with acute rejection. The scale is from 1 to 9, higher scores mean more severe signs of rejection.
Liver related complications | 24 months
  This endpoint will allow to assess the association between initial graft injury and liver specific complications in both study arms.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (2):
  - Rutgers New Jersey Medical School (New York), New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (2):
  - University Hospitals Leuven, Leuven
  - Institut de Recherche Expérimentale et Clinique (IREC) UCLouvain (Brussels), Woluwe-Saint-Lambert
- Institute for Clinical and Experimental Medicine (IKEM) (Prague), Prague, Czechia
- Copenhagen University Hospital, Copenhagen, Denmark
- Hôpital de la Croix-Rousse (Lyon), Lyon, France
- Germany (6):
  - Universitätsklinikum Essen, Essen
  - University Medical Centre Hamburg-Eppendorf, Hamburg-Eppendorf
  - Hannover Medical School, Hanover
  - University of Heidelberg, Heidelberg
  - University of Mainz, Mainz
  - University of Munich Grosshadern, München
- Italy (5):
  - Milano Institutio Nazionale dei Tumori (Milan), Milan
  - ASST Grande Ospedale Metropolitano Niguarda (Milan), Milan
  - Padova University Hospital, Padua
  - Gemelli University Hospital, Rome
  - University of Udine, Udine
- Lithuanian University of Health Sciences, Kaunas, Lithuania
- Netherlands (2):
  - University of Groningen and University Medical Centre Groningen, Groningen
  - University Medical Centre Rotterdam - Erasmus University Medical Center, Rotterdam
- Oslo University Hospital, Oslo, Norway
- Poland (2):
  - Department of Surgical Oncology, Transplant Surgery and General Surgery, Medical University of Gdańsk, Gdansk
  - Medical University of Warsaw, Warsaw
- Centro Hepato-Bilio-Pancreático e de Transplantação (CHBPT), Lisbon, Portugal
- Vall d'Hebron Barcelona Hospital Campus, Barcelona, Spain
- Karolinska Institutet (Stockholm), Stockholm, Sweden
- Switzerland (3):
  - Clarunis - University Digestive Health Care, Basel, Canton of Basel-City
  - University Hospital Zurich, Zurich, Canton of Zurich
  - Hôpitaux universitaires de Genève, Geneva
- United Kingdom (5):
  - University Hospitals Birmingham, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Royal Free Hospital (London), London
  - King's College Hospital (London), London
  - Freeman Hospital (Newcastle), Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eden J, Muller PC, Kuemmerli C, Peters F, Litke T, Kranich A, Kremer AE, von Felten S, Dutkowski P; HOPE4Cancer Trial Investigators. Hypothermic oxygenated perfusion (HOPE) against cancer recurrence after liver transplantation for hepatocellular carcinoma-study protocol for an international multicenter randomized controlled trial (HOPE4Cancer). Trials. 2025 Sep 26;26(1):369. doi: 10.1186/s13063-025-09120-1. PMID 41013675